CLINICAL TRIAL: NCT01971710
Title: Advancing Community Level Action for Improving MCH/PMTCT (ACCLAIM): A Multi-Country Randomized Trial to Evaluate the Effectiveness of Selected Community-Level Interventions on Key MCH/PMTCT Outcomes
Brief Title: Advancing Community Level Action for Improving MCH/PMTCT
Acronym: ACCLAIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Canadian International Development Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: EG112/113/115
Record Dates: First submitted 2013-08-13; First posted 2013-10-29 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: HIV
Keywords: HIV; AIDS; PMTCT
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Community Leader Engagement (Other): Trained formal and informal community leaders conducting community dialogues and advocacy, and developing community action plans
  Interventions: Behavioral: Community leader engagement
- Community Days (Other): Community gatherings involving participatory dialogue, guided discussion, and the provision of education and selected health services.
  Interventions: Behavioral: Community leader engagement; Behavioral: Community days
- Community Peer Groups (Other): Pregnant women attend 4 weekly peer-led classes in community peer groups. Men attending 4 peer-led education sessions in community peer groups
  Interventions: Behavioral: Community leader engagement; Behavioral: Community days; Behavioral: Community Peer Groups

INTERVENTIONS:
Behavioral: Community leader engagement — Community leaders conducting advocacy, community dialogue and community action plans on PMTCT/MCH
Behavioral: Community days — The provision of facilitated dialogues, advocacy and education, and selected health services, to a community on a specific day
  Arms: Community Days; Community Peer Groups
Behavioral: Community Peer Groups — Pregnant women in community peer groups receiving information and education on PMTCT/MCH through 4 weekly peer-led classes . Men in community peer groups receiving information and education on their role in supporting women and families through 4 peer-led education sessions.
  Arms: Community Peer Groups

SUMMARY:
The goal of the ACCLAIM (Advancing Community-Level Action for Improving MCH/PMTCT) project is to increase community demand for, uptake of, and retention in Maternal and Child Health (MCH) and/Prevention of Mother-to-child transmission of HIV (PMTCT) services to improve country progress toward elimination of pediatric HIV/AIDS.

DETAILED DESCRIPTION:
This study will undertake a three-arm randomized trial in Swaziland, Uganda and Zimbabwe. Districts/regions (n=9) with 45 PMTCT-implementing health facilities and their catchment areas (populations 7300-27500), will be randomly allocated to three intervention arms: 1) community leader engagement, 2) community leader engagement with community days, or 3) community leader engagement with community days and male and female community peer groups. The primary study outcome is HIV exposed infants (HEI) returning to the health facility within two months for early infant diagnosis (EID) of HIV. Secondary study outcomes include: gestational age of women attending for first antenatal care, male partners tested for HIV, and HEI receiving nevirapine prophylaxis at birth. Changes in community knowledge, attitudes, practices and beliefs on MCH/PMTCT will be assessed through household surveys.

ELIGIBILITY:
Inclusion Criteria:

* Must be a member of the community surveyed

Exclusion Criteria:

* Under 18 years of age

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 187335 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Proportion of HIV-exposed infants returning to health facility HIV testing | 6-8 weeks after birth
  The general objective for the study is to assess the efficacy of the three study arm activities on the uptake of, and retention of HIV positive pregnant/postpartum women in MCH/PMTCT services as measured by the proportion of infants returning to the health facility at 6-8 weeks of age for the early infant diagnosis (EID) of HIV.

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey Woelk, PhD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (3):
- Elizabeth Glaser Pediatric AIDS Foundation, Mbabane, Eswatini
- Elizabeth Glaser Pediatric AIDS Foundation, Kampala, Uganda
- Elizabeth Glaser Pediatric AIDS Foundation, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No
The dataset may be available in 2018. Enquiries may be made with the organization.

REFERENCES:
- [Derived] Woelk GB, Kieffer MP, Walker D, Mpofu D, Machekano R; Project ACCLAIM Study Group. Evaluating the effectiveness of selected community-level interventions on key maternal, child health, and prevention of mother-to-child transmission of HIV outcomes in three countries (the ACCLAIM Project): a study protocol for a randomized controlled trial. Trials. 2016 Feb 16;17:88. doi: 10.1186/s13063-016-1202-y. PMID 26883307